CLINICAL TRIAL: NCT01492686
Title: Efficacy and Safety Study of MCI-186 for Treatment of the Patients With Amyotrophic Lateral Sclerosis (ALS) 2
Brief Title: Phase 3 Study of MCI-186 for Treatment of Amyotrophic Lateral Sclerosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MCI186-19
Record Dates: First submitted 2011-12-11; First posted 2011-12-15 (Estimated); Results first posted 2018-12-31 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Amyotrophic Lateral Sclerosis (ALS)
Keywords: Amyotrophic Lateral Sclerosis (ALS)
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Edaravone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: MCI-186; Drug: MCI-186 in open label phase
- Arm 2 (Placebo Comparator)
  Interventions: Drug: Placebo; Drug: MCI-186 in open label phase

INTERVENTIONS:
Drug: MCI-186 — Two ampoules (60 mg) of MCI-186 injection are intravenously administered once a day, for successive 14 days, followed by 14 days observation period (first cycle). The following treatment (10 days' administration during 14 days) - observation (14 days) cycle is repeated five times (2nd-6th cycles).
  Arms: Arm 1
Drug: Placebo — Two ampoules of placebo injection are intravenously administered once a day, for successive 14 days, followed by 14 days observation period (first cycle). The following treatment (10 days' administration during 14 days) - observation (14 days) cycle is repeated five times (2nd-6th cycles).
  Arms: Arm 2
Drug: MCI-186 in open label phase — All patients after the double blind phase may receive MCI-186 in 7th until 12th treatment - observation cycles at the patients' will.

SUMMARY:
The primary objective of the study is to confirm the efficacy of 60 mg of MCI-186 via intravenous drip infusion once a day in the patients with ALS based on the changes in the revised ALS functional rating scale (ALSFRS-R) scores after 24 weeks administration in double-blind, placebo-controlled manner. The study is also to examine the safety of MCI-186 to the ALS patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients whose conditions are defined as "definite ALS"or "probable ALS"diagnostic criteria El Escorial and revised Airlie House.
* Patients who can eat a meal, excrete, or move with oneself alone, and do not need assistance in everyday life.
* Patients of less than 2 years after the onset of ALS.
* Patients whose progress of the condition during 12 weeks before administration meet other requirements.

Exclusion Criteria:

* Patients with such complications as Parkinson's disease, schizophrenia, dementia, renal failure, or other severe complication, and patients who have the anamnesis of hypersensitivity to edaravone.
* Pregnant, lactating, and probably pregnant patients, and patients who want to become pregnant, and patients who can not agree to contraception.
* Patients who have participated in other trials within 12 weeks before consent, or who are participating in other clinical trials at present.
* In addition to the above exclusion criteria, patients judged to be inadequate to participate in this study by their physician.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2011-12; Primary Completion 2014-09 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Osaka, Japan

REFERENCES:
- [Result] Writing Group; Edaravone (MCI-186) ALS 19 Study Group. Safety and efficacy of edaravone in well defined patients with amyotrophic lateral sclerosis: a randomised, double-blind, placebo-controlled trial. Lancet Neurol. 2017 Jul;16(7):505-512. doi: 10.1016/S1474-4422(17)30115-1. Epub 2017 May 15. PMID 28522181
- [Result] WRITING GROUP ON BEHALF OF THE EDARAVONE (MCI-186) ALS 19 STUDY GROUP. Open-label 24-week extension study of edaravone (MCI-186) in amyotrophic lateral sclerosis. Amyotroph Lateral Scler Frontotemporal Degener. 2017 Oct;18(sup1):55-63. doi: 10.1080/21678421.2017.1364269. PMID 28872920
- [Derived] Brooks BR, Pioro EP, Sakata T, Takahashi F, Hagan M, Apple S. The effects of intervention with intravenous edaravone in Study 19 on hospitalization, tracheostomy, ventilation, and death in patients with amyotrophic lateral sclerosis. Muscle Nerve. 2023 Oct;68(4):397-403. doi: 10.1002/mus.27946. Epub 2023 Jul 31. PMID 37525592
- [Derived] Takei K, Takahashi F, Liu S, Tsuda K, Palumbo J. Post-hoc analysis of randomised, placebo-controlled, double-blind study (MCI186-19) of edaravone (MCI-186) in amyotrophic lateral sclerosis. Amyotroph Lateral Scler Frontotemporal Degener. 2017 Oct;18(sup1):49-54. doi: 10.1080/21678421.2017.1361443. PMID 28872913

RESULTS

PARTICIPANT FLOW:
Groups:
- MCI-186: Double-blind MCI-186, Then Open-label MCI-186. 2 ampoules of edaravone injection 30 mg were administered once daily over 60 min by intravenous infusion.
- Placebo of MCI-186: Double-blind Placebo of MCI-186, Then Open-label MCI-186. 2 ampoules of edaravone injection placebo were administered once daily over 60 min by intravenous infusion.
Period: Double-blind Phase
Arm/Group | MCI-186 | Placebo of MCI-186
Started | 69 | 68
Completed | 67 | 60
Not Completed | 2 | 8
Not completed — Adverse Event | 0 | 2
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Due to a discontinuation criterion | 2 | 3
Period: Open-label Phase
Arm/Group | MCI-186 | Placebo of MCI-186
Started | 65 | 58
Completed | 53 | 40
Not Completed | 12 | 18
Not completed — Adverse Event | 1 | 2
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 6 | 7
Not completed — Due to a discontinuation criterion | 4 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MCI-186 | Placebo of MCI-186 | Total
Number analyzed (Participants) | 69 | 68 | 137
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 46 | 46 | 92
  >=65 years | 23 | 22 | 45
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 27 | 58
  Male | 38 | 41 | 79

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Revised ALS Functional Rating Scale (ALSFRS-R) Score in Full Analysis Set (FAS) Population at 24 Weeks
Description: 0=worst; 48=best
Time Frame: baseline and 24 weeks
Population: "1 patient who did not reach the end of cycle 3" was excluded from the FAS in the MCI-186 group.
  "2 patients who did not reach the end of cycle 3" were excluded from the FAS in the Placebo of MCI-186 group.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | MCI-186 | Placebo of MCI-186
Number analyzed (Participants) | 68 | 66
units on a scale | -5.01 (0.64) | -7.5 (0.66)

2. Secondary Outcome: Number of Participants With Death or a Specified State of Disease Progression
Description: Any of "death, disability of independent ambulation, loss of upper limbs function, tracheotomy, use of respirator, use of tube feeding and loss of useful speech" was defined as an event.
Time Frame: 24 weeks
Measure: Number; unit: Count of Participants
Arm/Group | MCI-186 | Placebo of MCI-186
Number analyzed (Participants) | 69 | 68
Count of Participants
  Death | 0 | 0
  Disability of independent ambulation | 0 | 2
  Loss of upper limbs function | 0 | 0
  Tracheotomy | 1 | 0
  Use of respirator | 0 | 0
  Use of tube feeding | 0 | 1
  Loss of useful speech | 1 | 3

3. Secondary Outcome: Change From Baseline in % Forced Vital Capacity (%FVC) in Full Analysis Set (FAS) Population at 24 Weeks
Time Frame: baseline and 24 weeks
Population: "1 patient who did not reach the end of cycle 3" and "1 patient with missing data" were excluded from the FAS in the MCI-186 group.
  "2 patients who did not reach the end of cycle 3" were excluded from the FAS in the Placebo of MCI-186 group.
Measure: Least Squares Mean (Standard Error); unit: percentage of FVC
Arm/Group | MCI-186 | Placebo of MCI-186
Number analyzed (Participants) | 67 | 66
percentage of FVC | -15.61 (2.41) | -20.4 (2.48)

4. Secondary Outcome: Change From Baseline in Modified Norris Scale Score in Full Analysis Set (FAS) Population at 24 Weeks
Description: The Modified Norris Scale is a measure of movement disorder for patients with ALS. 0=worst; 102=best
Time Frame: baseline and 24 weeks
Population: "1 patient who did not reach the end of cycle 3" was excluded from the FAS in the MCI-186 group.
  "2 patients who did not reach the end of cycle 3" and "3 patient with missing data" were excluded from the FAS in the Placebo of MCI-186 group.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | MCI-186 | Placebo of MCI-186
Number analyzed (Participants) | 68 | 63
units on a scale | -15.91 (1.97) | -20.8 (2.06)

5. Secondary Outcome: Change From Baseline in ALS Assessment Questionnaire (40 Items) (ALSAQ40) in Full Analysis Set (FAS) Population at 24 Weeks
Description: The ALSAQ40 score is a measure of QoL for patients with ALS. The ALSAQ40 evaluates domains that include physical mobility, Activities of daily living (ADL) and independence, eating and drinking, communication, and emotional reactions. 200=worst; 40=best
Time Frame: baseline and 24 weeks
Population: "1 patient who did not reach the end of cycle 3" was excluded from the FAS in the MCI-186 group.
  "2 patients who did not reach the end of cycle 3" and "2 patient with missing data" were excluded from the FAS in the Placebo of MCI-186 group.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | MCI-186 | Placebo of MCI-186
Number analyzed (Participants) | 68 | 64
units on a scale | 17.25 (3.39) | 26.04 (3.53)

6. Secondary Outcome: Percentage of Participants With Adverse Events
Time Frame: 24 weeks
Measure: Number; unit: percentage of Participants
Arm/Group | MCI-186 | Placebo of MCI-186
Number analyzed (Participants) | 69 | 68
percentage of Participants | 84.1 | 83.8

7. Secondary Outcome: Percentage of Participants With Adverse Drug Reactions
Time Frame: 24 weeks
Measure: Number; unit: percentage of Participants
Arm/Group | MCI-186 | Placebo of MCI-186
Number analyzed (Participants) | 69 | 68
percentage of Participants | 2.9 | 7.4

8. Secondary Outcome: Laboratory Tests Percentage of Participants With Adverse Events by System Organ Class (SOC) of "Investigations" (PT, MedDRA Ver. 17.0)
Time Frame: 24 weeks
Measure: Number; unit: percentage of Participants
Arm/Group | MCI-186 | Placebo of MCI-186
Number analyzed (Participants) | 69 | 68
percentage of Participants
  Blood bilirubin increased | 0 | 1.5
  Blood creatine phosphokinase increased | 0 | 1.5
  Liver function test abnormal | 1.4 | 1.5
  White blood cell count decreased | 1.4 | 0

9. Secondary Outcome: Percentage of Participants With Abnormal Values in Sensory Examinations
Time Frame: baseline and 24 weeks
Population: A note:
  Four patients of Placebo of MCI-186 group did not have data at 24 week. Therefore, concerning numbness (at 24 week) and staggering (at 24 week), the number of participants analysed are 64 in the both groups.
Measure: Number; unit: percentage of Participants
Arm/Group | MCI-186 | Placebo of MCI-186
Number analyzed (Participants) | 69 | 68
percentage of Participants
  Numbness (at baseline) | 2.9 | 7.4
  Numbness (at 24 week) | 7.2 | 9.4
  Staggering (at baseline) | 1.4 | 8.8
  Staggering (at 24 week) | 2.9 | 3.1

ADVERSE EVENTS:
Groups:
- Double-blind MCI-186: MCI-186 in Double-blind. 2 ampoules of edaravone injection 30 mg were administered once daily over 60 min by intravenous infusion.
- Double-blind Placebo of MCI-186: Placebo of MCI-186 in Double-blind. 2 ampoules of edaravone injection placebo were administered once daily over 60 min by intravenous infusion.
- Open-label MCI-186 (Double-blind MCI-186, Then Open-label): MCI-186 in Open-label (Double-blind MCI-186, Then Open-label). 2 ampoules of edaravone injection 30 mg were administered once daily over 60 min by intravenous infusion.
- Open-label MCI-186 (Double-blind Placebo, Then Open-label): MCI-186 in Open-label (Double-blind Placebo of MCI-186, Then Open-label). 2 ampoules of edaravone injection 30 mg were administered once daily over 60 min by intravenous infusion.
Arm/Group | Double-blind MCI-186 | Double-blind Placebo of MCI-186 | Open-label MCI-186 (Double-blind MCI-186, Then Open-label) | Open-label MCI-186 (Double-blind Placebo, Then Open-label)
Serious Adverse Events (participants affected / at risk) | 11/69 | 16/68 | 17/65 | 23/58
Other Adverse Events (participants affected / at risk) | 57/69 | 51/68 | 53/65 | 48/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Double-blind MCI-186 (N=69) | Double-blind Placebo of MCI-186 (N=68) | Open-label MCI-186 (Double-blind MCI-186, Then Open-label) (N=65) | Open-label MCI-186 (Double-blind Placebo, Then Open-label) (N=58)
Dysphagia (Gastrointestinal disorders) | 8 | 8 | 6 | 13
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Bacterial infection (Infections and infestations) | 1 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 0 | 1 | 3 | 2
Speech disorder (Nervous system disorders) | 1 | 2 | 2 | 1
Depression (Psychiatric disorders) | 0 | 1 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2 | 3
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 4 | 4
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0
Adjustment disorder (Psychiatric disorders) | 0 | 0 | 1 | 0
Stress cardiomyopathy (Cardiac disorders) | 0 | 0 | 0 | 1
Shock (Vascular disorders) | 0 | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 3
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Gait disturbance (General disorders) | 0 | 0 | 2 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Double-blind MCI-186 (N=69) | Double-blind Placebo of MCI-186 (N=68) | Open-label MCI-186 (Double-blind MCI-186, Then Open-label) (N=65) | Open-label MCI-186 (Double-blind Placebo, Then Open-label) (N=58)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Deafness neurosensory (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 1 | 0
Vertigo positional (Ear and labyrinth disorders) | 1 | 1 | 0 | 0
Blepharitis (Eye disorders) | 1 | 1 | 0 | 0
Eye discharge (Eye disorders) | 1 | 1 | 2 | 0
Retinal tear (Eye disorders) | 0 | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 2 | 0 | 0 | 1
Cheilitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 8 | 8 | 7 | 8
Diarrhoea (Gastrointestinal disorders) | 2 | 4 | 2 | 2
Dysphagia (Gastrointestinal disorders) | 0 | 2 | 6 | 13
Gastritis (Gastrointestinal disorders) | 1 | 0 | 3 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Malocclusion (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Periodontal disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 2
Catheter site dermatitis (General disorders) | 1 | 1 | 0 | 0
Feeling hot (General disorders) | 0 | 1 | 0 | 0
Infusion site erythema (General disorders) | 3 | 2 | 2 | 1
Infusion site pain (General disorders) | 3 | 2 | 0 | 1
Infusion site phlebitis (General disorders) | 0 | 1 | 0 | 0
Infusion site swelling (General disorders) | 0 | 2 | 1 | 0
Injection site rash (General disorders) | 0 | 1 | 0 | 0
Injection site reaction (General disorders) | 0 | 2 | 0 | 2
Pain (General disorders) | 0 | 1 | 1 | 2
Pyrexia (General disorders) | 0 | 3 | 1 | 0
Swelling (General disorders) | 1 | 0 | 0 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 2 | 0 | 0 | 1
Chronic sinusitis (Infections and infestations) | 1 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 1 | 0 | 0
Dermatitis infected (Infections and infestations) | 0 | 1 | 0 | 0
Device related infection (Infections and infestations) | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 1 | 2 | 0
Gingival abscess (Infections and infestations) | 1 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 1 | 0 | 1 | 0
Infected dermal cyst (Infections and infestations) | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 3 | 5 | 6 | 4
Oral herpes (Infections and infestations) | 0 | 1 | 0 | 0
Otitis externa (Infections and infestations) | 0 | 1 | 0 | 1
Periodontitis (Infections and infestations) | 1 | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 2 | 2 | 1 | 1
Postoperative wound infection (Infections and infestations) | 1 | 0 | 0 | 0
Tinea infection (Infections and infestations) | 1 | 0 | 0 | 0
Tinea pedis (Infections and infestations) | 1 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 1 | 1 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Chillblains (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 2
Contusion (Injury, poisoning and procedural complications) | 13 | 8 | 6 | 6
Excoriation (Injury, poisoning and procedural complications) | 2 | 2 | 3 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 2 | 1 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 2 | 2 | 1 | 2
Lip injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 1 | 4 | 2
Blood bilirubin increased (Investigations) | 0 | 1 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | 1 | 0
Liver function test abnormal (Investigations) | 1 | 1 | 0 | 0
White blood cell count decreased (Investigations) | 1 | 0 | 0 | 0
Gout (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 4 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 1 | 2 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 1 | 0 | 1
Myofascial pain syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1 | 1
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Carpal tunnel syndrome (Nervous system disorders) | 0 | 1 | 0 | 0
Decreased vibratory sense (Nervous system disorders) | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 2 | 2 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 4 | 5 | 1 | 3
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 1 | 0
Sciatica (Nervous system disorders) | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 5 | 4 | 2 | 2
Dysuria (Renal and urinary disorders) | 1 | 0 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 2 | 2 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 4 | 4
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 5 | 2 | 4 | 1
Asteatosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 8 | 3 | 3 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 5 | 2 | 5 | 2
Erythema (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Henoch-Schonlein purpura (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0
Miliaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 3 | 5 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 2 | 1 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 1
Hypertension (Vascular disorders) | 1 | 0 | 1 | 1
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0
Phlebitis (Vascular disorders) | 0 | 2 | 0 | 0
Vasculitis (Vascular disorders) | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0
Gingivitis (Infections and infestations) | 0 | 0 | 0 | 1
Herpes simplex (Infections and infestations) | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 1 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 1
Tinea cruris (Infections and infestations) | 0 | 0 | 1 | 0
Catheter site infection (Infections and infestations) | 0 | 0 | 2 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 1 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 0 | 1
Neurosis (Psychiatric disorders) | 0 | 0 | 1 | 0
Adjustment disorder (Psychiatric disorders) | 0 | 0 | 1 | 0
Speech disorder (Nervous system disorders) | 0 | 0 | 2 | 1
Tremor (Nervous system disorders) | 0 | 0 | 1 | 0
Conjunctivitis allergic (Eye disorders) | 0 | 0 | 1 | 0
Diplopia (Eye disorders) | 0 | 0 | 0 | 1
Dry eye (Eye disorders) | 0 | 0 | 1 | 0
Eczema eyelids (Eye disorders) | 0 | 0 | 1 | 0
Sudden hearing loss (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Stress cardiomyopathy (Cardiac disorders) | 0 | 0 | 0 | 1
Shock (Vascular disorders) | 0 | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 3
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 3
Change of bowel habit (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Dental caries (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Anal inflammation (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Epigastric discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Excessive granulation tissue (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 2
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 2
Tendon pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 1 | 0
Incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 1
Nocturia (Renal and urinary disorders) | 0 | 0 | 1 | 0
Gait disturbance (General disorders) | 0 | 0 | 2 | 0
Malaise (General disorders) | 0 | 0 | 1 | 0
Catheter site haemorrhage (General disorders) | 0 | 0 | 1 | 1
Catheter site erythema (General disorders) | 0 | 0 | 0 | 1
Catheter site inflammation (General disorders) | 0 | 0 | 1 | 0
Infusion site pruritus (General disorders) | 0 | 0 | 1 | 0
Puncture site swelling (General disorders) | 0 | 0 | 0 | 1
Blood pressure increased (Investigations) | 0 | 0 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 1
Blood urine present (Investigations) | 0 | 0 | 0 | 1
White blood cell count increased (Investigations) | 0 | 0 | 1 | 0
Protein urine present (Investigations) | 0 | 0 | 0 | 1
Bite (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Wound compliation (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other